CLINICAL TRIAL: NCT05867459
Title: Maternal and Fetal Outcome of CKD Mother Patient in Sohag Governorate
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamd Saad Mohamedein, internal medicine resident in sohag university hospital, Sohag University
Other Study IDs: Soh-Med-23-04-06MS
Record Dates: First submitted 2023-05-02; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: CKD PREGNANT WOMEN
MeSH Terms: interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD PREGNANT PATIENT: The Group of pregnant CKD PT as mentioned in introduction and according to KIDOG definition of CKD regardless cause of CKD
  Interventions: Diagnostic Test: Serum creatinine; Diagnostic Test: Alb /creat ratio or 24h urine protein; Diagnostic Test: Serum electrolyte; Diagnostic Test: Urine analysis; Diagnostic Test: Abdominal ultrasound; Diagnostic Test: Renal biobsy; Other: Clinical assesment

INTERVENTIONS:
Diagnostic Test: Serum creatinine — The test wil be measured for all pt in study to detect of their grade of CKD
Diagnostic Test: Alb /creat ratio or 24h urine protein — Test will be measured to detect type and sevirity of proteinuria
Diagnostic Test: Serum electrolyte — The test will be measured in all pt to detect renal tubular state
Diagnostic Test: Urine analysis — It is mirror of kidney
Diagnostic Test: Abdominal ultrasound — To detect the anatomy and any structural abnormality in kidneys
Diagnostic Test: Renal biobsy — Is done but not for all pt but for pt that can do it and agree for it .the test is used for detection of type of CKD or type of glomerionephritis
Other: Clinical assesment — Clinical assessment:
  age, kidney disease history, history of DM or HTN ,history of pregnancy during study, therapy in early pregnancy , body weight, body height, and . Mean arterial pressure (MAP) . Body mass index (BMI). According to age and Scr level, the estimated glomerular filtration rate (eGFR) was calculated by CKD-EPI Creatinine Equation (2021)
  Evaluation of pregnancy outcomes :Adverse pregnancy outcomes included maternal death, severe preeclampsia ,eclampsia ,duration of hospital stay and type of care need, mode of delivery ,need of blood transfusion , gestational age during delivary for detet preterm birth early preterm or late preterm from or extremely preterm > 28W, birth weigh for low birthweight ,very low birth weight , extremely low birth weight,NICU admission,IUGR, still birth ,abortion, and neonatal death.

SUMMARY:
Aim of the work:

In this study, we aimed:

Is to investigate the following issues: (1) the pregnancy outcomes of patients with CKD (2) additional risk factors for adverse pregnancy outcomes in patients with CKD in the area of sohag governorate.

DETAILED DESCRIPTION:
prospective observational study including group of pregnant CKD women The Group of pregnant CKD PT as mentioned in introduction and according to KIDOG definition of CKD regardless cause of CKD .

The data will be collected by multiple visit and survey of patient in hemodialysis units in sohag governorate and renal outpatient clinic and obstetric department and internal medicine department in sohag university hospital

Duration of study:

nine month after approval of protocol by medical research committee of sohag faculty of medicine

Data collection procedure:

The following clinical data will be collected:

Clinical assessment:

age, kidney disease history, history of DM or HTN ,history of pregnancy during study, therapy in early pregnancy (including antihypertensive drugs and immunosuppressive agents), , baseline blood pressure, body weight, body height, and . Mean arterial pressure (MAP) was calculated as (systolic pressure+2×diastolic pressure)/3. Body mass index (BMI) was calculated based on height and body weight. According to age and Scr level, the estimated glomerular filtration rate (eGFR) was calculated by CKD-EPI Creatinine Equation (2021)

Evaluation of pregnancy outcomes :Adverse pregnancy outcomes included maternal death, severe preeclampsia ,eclampsia ,duration of hospital stay and type of care need, mode of delivery ,need of blood transfusion , gestational age during delivary for detet preterm birth> 37W early preterm from 28 to 34W or late preterm from 34 to37W or extremely preterm > 28W, birth weigh for low birthweight> 2500 g ,very low birth weight >1500g , extremely low birth weight>1000g,NICU admission,IUGR, still birth ,abortion, and neonatal death.

Laboratory assessment:

1. serum creatinine
2. urine analysis 3-24h protein in urine or albumin create ratio

4-serum electrolyte s.Na s.K ionezed Ca 5-pathological result of renal biopsy if done 6-abdominal ultrasound with full comment on kidney

ELIGIBILITY:
Inclusion Criteria:

* All pregnant patients with CKD regardless the cause of CKD in any stage of CKD on dialysis or not.

Exclusion Criteria:

* Any patient not defined CKD or serum creatinineless than1,2 befor 13W of pregnancy Grand multipara patient with history of multiple abortion or still birth not related to CKD affection period

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any patient in hemodialysis units in sohag governorate and renal outpatient clinic and obstetric department and internal medicine department in sohag university hospital has the crietria of CKD pregnant women
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
1) the pregnancy outcomes of patients with CKD (2) additional risk factors for adverse pregnancy outcomes in patients with CKD | From day of enrollment of pt in study to one week after delivary
  Medical and clinial data will collect And retrospectively analyze. The data well collected by multiple visit to pt or telephon calling for follow up data will ensured by report of about pt from obstetric and nicu doctor Evaluation of pregnancy outcomes :Adverse pregnancy outcomes included maternal death, severe preeclampsia ,eclampsia The diagnostic criteria for severe preeclampsia were based on the 2013 Hypertension in Pregnancy Guidelines of the American College of Obstetricians and Gynecologists .
  duration of hospital stay and type of care need, mode of delivery ,need of blood transfusion , gestational age during delivary for detet preterm birth and its type, birth weigh for detect low birth Wt and its degree ,NICU admission,IUGR as fetus is 10 centile according gastational age, still birth, ,abortion , and neonatal death, any documented congenital anomalies of fetus.
  And questionaire of pt for risk factor as DM,HTN,maternal age,drug use during delivary, stage of CKD

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cabiddu G, Castellino S, Gernone G, Santoro D, Moroni G, Giannattasio M, Gregorini G, Giacchino F, Attini R, Loi V, Limardo M, Gammaro L, Todros T, Piccoli GB. A best practice position statement on pregnancy in chronic kidney disease: the Italian Study Group on Kidney and Pregnancy. J Nephrol. 2016 Jun;29(3):277-303. doi: 10.1007/s40620-016-0285-6. Epub 2016 Mar 17. PMID 26988973
- [Background] Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, Kusek JW, Van Lente F; Chronic Kidney Disease Epidemiology Collaboration. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Ann Intern Med. 2006 Aug 15;145(4):247-54. doi: 10.7326/0003-4819-145-4-200608150-00004. PMID 16908915
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Result] Hall M. Pregnancy in Women With CKD: A Success Story. Am J Kidney Dis. 2016 Oct;68(4):633-639. doi: 10.1053/j.ajkd.2016.04.022. Epub 2016 Jun 25. PMID 27350132